CLINICAL TRIAL: NCT00674297
Title: Effects of Fluvastatin on Proinflammatory and Prothrombotic Markers in Antiphospholipid Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 28005
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Antiphospholipid Syndrome
Keywords: Persistently Antiphospholipid Antibody Positive Patients
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluvastatin (Experimental): All patients will take Fluvastatin 40 mg daily for 3 months.
  Interventions: Drug: Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin — Fluvastatin 40 mg daily for 3 months
  Other Names: Lescol, Lescol XL

SUMMARY:
The purpose of this study is to determine whether a drug named Fluvastatin is beneficial and safe in reducing the risk of cardiovascular disease and blood clots in patients with antiphospholipid antibodies or Antiphospholipid Syndrome (APS).

DETAILED DESCRIPTION:
The primary objective of the study is to determine the effects of fluvastatin on pro-thrombotic and pro-inflammatory markers in aPL-positive lupus and non-lupus patients (primary endpoint) and to determine the safety of fluvastatin in aPL-positive lupus and non-lupus patients (secondary endpoint).

All eligible patients will sign an IRB-approved consent form during the screening visit and give blood for baseline laboratory tests. Within a week of the screening visit, all patients will be started on Fluvastatin 40 mg daily for three months. At three months patients will be instructed to stop the study medication and they will be followed for another three months. Thus, the total duration of the study is six months: first three months is interventional and the last three months is observational.

ELIGIBILITY:
Inclusion Criteria:

* Persistently antiphospholipid-antibody positive patients (positive lupus anticoagulant test, anticardiolipin antibody ≥ 40 GPL /MPL, and/or anti- β2-glycoprotein I antibody > 20 SGU/SMU) with or without systemic lupus erythematosus

Exclusion Criteria:

* Younger than 18 year-old
* Pregnant
* Planning to get pregnant within the next 6 months
* Taking other cholesterol lowering agents
* Taking other immunosuppressive medications (such as methotrexate, azathioprine, cellcept, enbrel, remicade, or rituximab)(Hydroxychloroquine [Plaquenil] during the study period is allowed).
* Treatment with biologic agents including anti-TNF medications and Rituximab
* Treatment with erythromycin, itraconazole, or clarithromycin
* Taking prednisone higher than 10 mg daily
* Taking non-steroidal anti-inflammatory drug (such as Motrin, Advil, etc) regularly
* Have a muscle or liver disease
* Have chronic renal disease requiring dialysis
* Have hepatitis C and/or HIV infection
* Have active infections requiring antibiotics
* Have the diagnosis of a systemic autoimmune disease (such as rheumatoid arthritis or systemic sclerosis) other than lupus
* Have diagnosis of another chronic condition requiring corticosteroid treatment more than 10mg daily
* History of an allergic reaction to cholesterol lowering agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doruk Erkan, MD, Principal Investigator — Hospital for Special Surgery, New York; Silvia Pierangeli, PhD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - Division of Rheumatology, University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erkan D, Willis R, Murthy VL, Basra G, Vega J, Ruiz-Limon P, Carrera AL, Papalardo E, Martinez-Martinez LA, Gonzalez EB, Pierangeli SS. A prospective open-label pilot study of fluvastatin on proinflammatory and prothrombotic biomarkers in antiphospholipid antibody positive patients. Ann Rheum Dis. 2014 Jun;73(6):1176-80. doi: 10.1136/annrheumdis-2013-203622. Epub 2013 Aug 9. PMID 23933625
- See also: A prospective open-label pilot study of fluvastatin on proinflammatory and prothrombotic biomarkers in antiphospholipid antibody positive patients — http://www.ncbi.nlm.nih.gov/pubmed/23933625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 groups were recruited: primary antiphospholipid syndrome(PAPS); systemic lupus erythematosus (SLE) with antiphospholipid syndrome(APS)(SLE/APS); persistent aPL positivity without SLE/APS(Primary aPL); and persistent aPL positivity with SLE but no APS(SLE/ aPL). The frequency-matched control group was identified from a databank of healthy persons.
Pre-assignment Details: SLE was defined based on the American College of Rheumatology classification criteria. APS was defined based on the updated Sapporo classification criteria.
  Positive aPL was defined as persistently (at least 12 weeks apart) positive LA test, aCL≥40 GPL/MPL and/or aβ2GPI≥20 SGU/SMU.
Groups:
- PAPS: Primary APS
- SLE/APS: SLE with APS
- Primary aPL: Persistant aPL positivity without SLE or APS.
- SLE/aPL: Persistent aPL positivity with SLE but no APS.
Period: Overall Study
Arm/Group | PAPS | SLE/APS | Primary aPL | SLE/aPL
Started (41 patients recruited.) | 18 | 7 | 9 | 7
Completed (24 patients completed the study.) | 8 | 7 | 5 | 4
Not Completed | 10 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Arm/Group | Fluvastatin
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants] — Ages between 18 and 65
  Participants
    <=18 years | 0
    Between 18 and 65 years | 41
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 28
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Effects of Fluvastatin on Proinflammatory and Prothrombotic Biomarkers (BMR) in aPL Positive Patients
Description: Biomarkers: IL6 (pg/mL), IL1β (pg/mL), IL8 (pg/mL), VEGF (pg/mL), TNFα (pg/mL), IFNα (pg/mL), IP10 (pg/mL), sCD40L (pg/mL)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PAPS | SLE/APS | Primary aPL | SLE/aPL
Number analyzed (Participants) | 18 | 7 | 9 | 7
pg/mL
  Biomarker IL6 | 31.2 (48.4) | 12.2 (103.5) | 0.4 (0.7) | 2.7 (76.8)
  Biomarker IL1B | 3.0 (7.7) | 11.4 (20.1) | 0.3 (0.6) | 0.5 (5.1)
  Biomarker IL8 | 24.5 (48.4) | 27.4 (53.7) | 7.2 (50.4) | 21.6 (48.9)
  Biomarker VEGF | 242.2 (399.6) | 109.1 (348.4) | 74.6 (158.3) | 67.2 (499.4)
  Biomarker TNFa | 21.5 (50.5) | 11.6 (24.1) | 8.9 (15.7) | 53.9 (62.5)
  Biomarker IFNa | 10.1 (88.4) | 0.3 (367.1) | 0.3 (512.2) | 13.2 (558.5)
  Biomarker IP10 | 427.2 (569.8) | 656.2 (454.8) | 249.7 (698.9) | 472.5 (690.5)
  Biomarker sCD40L | 276.5 (676.0) | 145.6 (5159.8) | 149.7 (17035.6) | 76.9 (970.0)

2. Primary Outcome: Effects of Fluvastatin on Proinflammatory and Prothrombotic Biomarkers (BMR) in aPL Positive Patients
Description: Biomarker sTF (pM)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pM
Arm/Group | PAPS | SLE/APS | Primary aPL | SLE/aPL
Number analyzed (Participants) | 18 | 7 | 9 | 7
pM | 153.6 (381.0) | 329.2 (447.0) | 190.4 (139.0) | 102.1 (177.0)

3. Primary Outcome: Effects of Fluvastatin on Proinflammatory and Prothrombotic Biomarkers (BMR) in aPL Positive Patients
Description: Biomarkers sICAM-1 (ng/mL), sVCAM-1 (ng/mL), sE-sel (ng/mL)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PAPS | SLE/APS | Primary aPL | SLE/aPL
Number analyzed (Participants) | 18 | 7 | 9 | 7
ng/mL
  sICAM-1 | 281.6 (406.8) | 55.1 (70.3) | 163.5 (341.7) | 2.8 (32.9)
  sVCAM-1 | 1128.4 (1152.8) | 156.4 (19.3) | 321.3 (1015.1) | 41.1 (27.2)
  sE-sel | 27.7 (36.7) | 14.7 (20.4) | 10.9 (26.4) | 4.1 (21.5)

ADVERSE EVENTS:
Time Frame: 6 months
Description: An adverse event (AE) was defined as any untoward medical occurrence in a study patient regardless of causality assessment. A serious AE was defined as one occurring at any dose that met one or more of the following criteria: death; life-threatening; requiring or prolonging inpatient hospitalisation; disabling; or resulting in a congenital anomaly/birth defect.
Groups:
- aPL Positive Patients: Patients with aPL positivity
Arm/Group | aPL Positive Patients
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 8/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aPL Positive Patients (N=41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lupus flare (Immune system disorders) | 1 (1)
Myalgia with high CPK (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia with normal CPK (Musculoskeletal and connective tissue disorders) | 3 (3)
Recurrent deep vein thrombosis (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No